CLINICAL TRIAL: NCT03858322
Title: 'ADVANCE' (A Pilot Trial) ADjuVANt Chemotherapy in the Elderly: Developing and Evaluating Lower-Toxicity Chemotherapy Options for Older Patients With Breast Cancer
Brief Title: 'ADVANCE' (A Pilot Trial)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Rachel Freedman, MD, MPH, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-031
Record Dates: First submitted 2019-02-25; First posted 2019-02-28 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Cyclophosphamide; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Carboplatin + Paclitaxel (Experimental): * Paclitaxel will be administered intravenously 3 times per cycle
  * Carboplatin will be administered intravenously 3 times per cycle
  Interventions: Drug: Paclitaxel; Drug: Carboplatin
- Cyclophosphamide + Paclitaxel (Experimental): * Paclitaxel will be administered intravenously 3 times per cycle
  * Cyclophosphamide will be administered once per cycle
  Interventions: Drug: Paclitaxel; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Paclitaxel — The drug work by damaging the RNA or DNA that tells the cell how to copy itself in division. If the cells are unable to divide, they die.
Drug: Cyclophosphamide — The drug work by damaging the RNA or DNA that tells the cell how to copy itself in division. If the cells are unable to divide, they die.
  Arms: Cyclophosphamide + Paclitaxel
Drug: Carboplatin — The drug work by damaging the RNA or DNA that tells the cell how to copy itself in division. If the cells are unable to divide, they die.
  Arms: Carboplatin + Paclitaxel

SUMMARY:
This study is being conducted to carefully study how chemotherapy is tolerated in group of patients age 70.

DETAILED DESCRIPTION:
This clinical trial is dedicated to patients age 70 and older and is focused on understanding how the investigators can improve upon breast cancer outcomes for older women, a group of patients who often do worse than younger patients and who are not well represented in clinical trials to date. Through this clinical trial, the investigators aim to better understand the side effects, experiences, and changes in physical function that may occur with chemotherapy. The investigators are also very interested in the genomics (or gene-changes) and biological changes that may occur in breast cancers in older women that may be different from the changes we see in younger patients.

Even though the chemotherapy agents being used in this study are used frequently when treating breast cancer, The investigators have limited information on how these agents are tolerated in older patients. This research study is called a Feasibility Study, because the investigators will be closely monitoring how easily it is to administer chemotherapy to a relatively small group of participants (up to 40) and to what degree side effects occur. The investigators will administer commercially available chemotherapy agents used in breast cancer in the specific setting of the treating older patients with early-stage breast cancer and with some mild modification of how these agents are given and in what combination.

For participants with triple negative breast cancer, paclitaxel and carboplatin will be administered in standard, weekly doses. Both agents are FDA-approved for use in early breast cancer. However, carboplatin and paclitaxel are not typically used as a 'stand-alone' treatment for breast cancer, meaning they are often used together along with other chemotherapy agent(s) over a longer period.

For participants with hormone receptor-positive breast cancer, paclitaxel and cyclophosphamide will be administered, which are both FDA-approved agents to treat breast cancer as part of a longer regimen to treat early breast cancer. In this clinical trial the investigators are modifying the way the chemotherapy is delivered so that it may be more tolerable than the longer treatment course. This clinical trial does not limit the use of other chemotherapy or other treatments being recommended for breast cancer, but any other recommended treatments would be given after the participants receive their paclitaxel and carboplatin on the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed breast cancer that is human epidermal growth factor receptor 2 negative (HER2-negative) per the most recent 2018 ASCO CAP guidelines94
* Estrogen Receptor and Progesterone immunohistochemistry (IHC) status must be known; any status is eligible, but this will define in which cohort a patient will enroll:
* Additional eligibility for cohort 1: Triple negative disease- defined as IHC staining of <10% for ER and PR per local pathology review
* Additional eligibility for cohort 2: Hormone receptor-positive disease defined as IHC for ER or PR >/= 10% per local pathology review
* Men and women are eligible
* Age 70 and older at the time of protocol registration
* Non-metastatic, invasive breast cancer (scans are not required to document non-metastatic disease- any staging work-up is up to the treating provider's discretion)
* Recommended to have either neoadjuvant chemotherapy or adjuvant chemotherapy per their treating provider.
* Any surgery, nodal assessment, radiation, hormonal therapy is left up to the treating provider but should not occur concurrently with study therapy. If any additional chemotherapy is planned by a treating provider, this must occur AFTER all study-related chemotherapy is completed.
* Any patient receiving pre-operative hormonal therapy and who is then recommended for adjuvant chemotherapy is eligible, though hormonal therapy should be held during study treatment administration
* All study-related chemotherapy must be given prior to surgery if neoadjuvant therapy is planned or adjuvantly if postoperative chemotherapy is planned. For example, giving 6 doses pre-operatively and 6 doses postoperatively is not allowed on study.
* There are no restrictions on life expectancy, ECOG Performance Status, or baseline blood values or organ function; Appropriateness of chemotherapy treatment is left up to the treating provider but providers should be ok with the full starting doses of each agent.
* Participants must be willing to fill out surveys over time or designate a proxy to answer on their behalf.
* Ability to understand and the willingness to sign a written informed consent document.
* Patients who do not speak or read English are eligible as long as adequate interpreter services are available or the surveys are available in the preferred language (i.e. PRO surveys are available in many languages)

Exclusion Criteria:

* Participants who have already received chemotherapy for the current cancer. Prior diagnoses of breast cancers are allowed, provided that the treating provider feels that the current cancer represents a new primary breast cancer and not recurrent disease.
* Participants who are receiving any other investigational or anti-cancer agents. Any additional radiation, hormonal therapy or chemotherapy planned should be administered once the study treatments have completed.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cyclophosphamide, carboplatin, and paclitaxel.
* Prior chemotherapy receipt is allowed in the setting of treatment of other/prior cancers, but no prior carboplatin (cohort 1), cyclophosphamide (cohort 2), or paclitaxel (both cohorts) receipt in the last 2 years is allowed (given toxicity and possible efficacy concerns

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2019-03-21 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Toxicity and receipt of planned therapy (feasibility) | 3 months
  Examine the number of treatments received divided by the denominator of 12 treatments

SECONDARY OUTCOMES:
Adverse events | 2 years
  Using CTCAE standard reporting
NCI PRO-CTCAE | 2 Years
  Examine patient reported CTCAEs on study treatment and their agreement with provider reports.
Consequences of toxicity or disease events | 2 years
  Frequency of hospitalizations, deaths, emergency room visits
Invasive disease-free survival | 2 years
  recurrences and survival as per STEEP definitions and whether recurrences are local or distant
Overall survival | 2 years
  We will examine the time from study registration to death

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Freedman, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (5):
- United States (5):
  - City of Hope National Medical Center, Duarte, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center (DF/BWCC) at Milford Regional Medical Center, Milford, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center (DF/BWCC) in Clinical Affiliation with South Shore Hospital, South Weymouth, Massachusetts
  - Novant Health Oncology Specialists, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: BCH - Contact the Technology & Innovation Development Office at www.childrensinnovations.org or email TIDO@childrens.harvard.edu BIDMC - Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu BWH - Contact the Partners Innovations team at http://www.partners.org/innovation DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu MGH - Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Derived] Mayerhofer C, Sedrak MS, Hopkins JO, Li T, Tayob N, Faggen MG, Sinclair NF, Chen WY, Parsons HA, Mayer EL, Lange PB, Basta AS, Perilla-Glen A, Lederman RI, Wong AR, Tiwari A, McAllister SS, Mittendorf EA, Gibson CJ, Burstein HJ, Kim AS, Freedman RA, Miller PG. Clonal hematopoiesis in older patients with breast cancer receiving chemotherapy. J Natl Cancer Inst. 2023 Aug 8;115(8):981-988. doi: 10.1093/jnci/djad065. PMID 37042724
- [Derived] Freedman RA, Li T, Sedrak MS, Hopkins JO, Tayob N, Faggen MG, Sinclair NF, Chen WY, Parsons HA, Mayer EL, Lange PB, Basta AS, Perilla-Glen A, Lederman RI, Wong A, Tiwari A, McAllister SS, Mittendorf EA, Miller PG, Gibson CJ, Burstein HJ. 'ADVANCE' (a pilot trial) ADjuVANt chemotherapy in the elderly: Developing and evaluating lower-toxicity chemotherapy options for older patients with breast cancer. J Geriatr Oncol. 2023 Jan;14(1):101377. doi: 10.1016/j.jgo.2022.09.006. Epub 2022 Sep 23. PMID 36163163

DOCUMENTS (1):
  • Informed Consent Form (2020-02-26): https://cdn.clinicaltrials.gov/large-docs/22/NCT03858322/ICF_000.pdf